CLINICAL TRIAL: NCT03625024
Title: Quality Assurance of Cognitive-behavioral Therapy: Adherence and Competence in Therapists and Treatment Outcome in Patients With Depression and Anxiety
Brief Title: Quality Assurance of Cognitive-behavioral Therapy
Status: Completed | Type: Observational
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Benjamin Bohman, Associate professor, Karolinska Institutet
Other Study IDs: KI-2018/472-31/5
Record Dates: First submitted 2018-06-28; First posted 2018-08-10 (Actual); Last update posted 2022-08-26 (Actual); Status verified 2022-08

CONDITIONS: Depression, Anxiety
MeSH Terms: conditions — Depression; Anxiety Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Cognitive-behavioral therapy — Individual cognitive-behavioral therapy, including homework and behavioral change methods.

SUMMARY:
The study examines associations between competence in cognitive-behavioral therapy (CBT) and adherence to evidence-based generic CBT in therapists and treatment outcome in patients with depression or an anxiety disorder in psychiatric outpatient care.

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of major depression or an anxiety disorder (panic disorder, agoraphobia, social anxiety, generalized anxiety disorder, obsessive-compulsive disorder, post-traumatic stress disorder)

Exclusion Criteria:

* Psychosis, bipolar disorder, eating disorder, substance use disorder, high risk of suicide, any simultaneous psychological treatment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients in psychiatric outpatient care with depression or anxiety disorder.
Sampling Method: Non-Probability Sample
Enrollment: 89 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2021-11-22 (Actual); Study Completion 2021-11-22 (Actual)

PRIMARY OUTCOMES:
Disorder-specific self-reported symptoms change instruments | Change from baseline symptoms at 18 weeks
  Symptoms measures of depression or an anxiety disorder

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Bohman, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- WeMind Psykiatri, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bergvall H, Linde J, Alfonsson S, Sunnhed R, Barber JP, Lundgren T, Andersson G, Bohman B. Quality of cognitive-behavioural therapy in routine psychiatric care: therapist adherence and competence, and patient outcomes for depression and anxiety disorders. BMC Psychiatry. 2024 Dec 4;24(1):887. doi: 10.1186/s12888-024-06328-4. PMID 39633319